CLINICAL TRIAL: NCT03585439
Title: Isthmic Spondylolisthesis Treated With Circumferential Arthrodesis Combining Anterior Lumbar Interbody Fusion With Posterolateral Fusion. About 150 Cases
Brief Title: Isthmic Spondylolisthesis Treated With Combined Approach: Clinical and Radiological Outcomes
Acronym: SPLAC
Status: Completed | Type: Observational
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/06
Record Dates: First submitted 2018-06-06; First posted 2018-07-13 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Isthmic Spondylolisthesis; Surgical Procedure, Unspecified
Keywords: Isthmic spondylolisthesis; vertebral fusion; combined approach; circumferential fusion; ALIF; posterior fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single cohort of operated patients: One group of patients: isthmic spondylolisthesis operated in our center using a double approach technique
  Interventions: Procedure: Observational study evaluating the results of an intervention for isthmic spondylolisthesis: surgical procedure with double approach: Anterior lumbar Interbody Fusion then postero-lateral fusion

INTERVENTIONS:
Procedure: Observational study evaluating the results of an intervention for isthmic spondylolisthesis: surgical procedure with double approach: Anterior lumbar Interbody Fusion then postero-lateral fusion — First in supine position, an ALIF is performed: with a Pfannenstiel incision, through a retroperitoneal approach, a discectomy is performed at the level of the spondylolisthesis then a cage is placed between the two vertebral bodies. Then, in prone position, a standard posterior approach is performed, pedicle screws are placed to achieve a postero-lateral fusion. A decompression may be associated.

SUMMARY:
This study aims to evaluate clinical and radiological outcomes of isthmic spondylolisthesis surgically treated with combined approach. The goal is to demonstrate that it is a safe and efficient technique to treat isthmic spondylolisthesis. There is very little literature concerning this procedure.

DETAILED DESCRIPTION:
Isthmic spondylolisthesis can cause back and leg pain. If pain persists after well conducted medical management, a surgical treatment can be proposed. Even though the goal is consensual, there are plenty of ways to reach vertebral fusion: ALIF, PLIF, TLIF, Posterior fusion only, etc… This study aims to evaluate clinical and radiological outcomes of isthmic spondylolisthesis surgically treated with combined approach. The goal is to demonstrate that it is a safe and efficient technique to treat isthmic spondylolisthesis using standard XRays, CT Scan and patient reported outcome measurements. There is very little literature concerning this procedure.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged over 18 years
* With isthmic spondylolisthesis at L4-L5 or L5-S1
* Operated in our center with a double approach: Anterior lumbar interbody fusion then postero-lateral fusion
* Consent for participation

Exclusion Criteria:

* Pseudarthrosis L5-S1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive cohort of patients operated in our center from 2013 to 2017
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Fusion status | From 6 months to 1 year after surgery
  Every patient has a CT-Scan of the lumbar spine done to check fusion status. The interpretation is made by the surgeon who did the surgery and one independent reviewer.

SECONDARY OUTCOMES:
Restoration of the foraminal diameter | 3 months and 1 year after surgery
  The foraminal diameter is measured to quantify the restoration of the foraminal diameter after surgery, making more room for the nerve root.
Correction of the spondylolisthesis-induced kyphosis after surgery | 3 months and 1 year after surgery
  The lumbo-sacral angle is measured to quantify the correction of the spondylolisthesis-induced kyphosis after surgery.
Segmental lordosis | 3 months and 1 year after surgery
  Segmental lordosis is measured with the L5-S1 lordosis, quantifying the correction at the spondylolisthesis level
Local Lordosis | 3 months and 1 year after surgery
  Local Lordosis measured with the L4-S1 lordosis, quantifying the correction in the lower lumbar region
Back pain | Pre-operative, 3 months and 1 year after surgery
  Measured with Lumbar Visual Analogic Scale. The patient quantifies his back pain with a number, ranging from 0 to 10 (0 = no pain, 10= worst possible pain)
Sciatica | Pre-operative, 3 months and 1 year after surgery
  Measured with Radicular Visual Analogic Scale. The patient quantifies his leg pain with a number, ranging from 0 to 10 (0 = no pain, 10= worst possible pain)
Disability | Pre-operative, 3 months and 1 year after surgery
  Measured with the ODI (Oswestry Disability Index). The patient answers 10 questions concerning his daily life and the disability caused by his back problem, giving a global score. 0 is equated with no disability and 100 is the maximum disability possible.
Complication rate | until 1 year after surgery
  intra-operative, early and late post-operative complications (vascular injury, non-union, infection, etc…)

CONTACTS AND LOCATIONS:
Locations (1):
- CMC Ambroise Pare, Neuilly-sur-Seine, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No